CLINICAL TRIAL: NCT01959698
Title: Phase I/Ib Study of Carfilzomib Plus Rituximab Plus Ifosfamide Plus Carboplatin Plus Etoposide (C-R-ICE) in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Carfilzomib, Rituximab, Ifosfamide, Carboplatin, and Etoposide in Treating Patients With Relapsed or Refractory Stage I-IV Diffuse Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 240813; NCI-2013-01784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 240813 (Other: Roswell Park Cancer Institute); R01CA136907 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: CD20 Positive; Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Stage I Diffuse Large B-Cell Lymphoma; Stage II Diffuse Large B-Cell Lymphoma; Stage III Diffuse Large B-Cell Lymphoma; Stage IV Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Carboplatin; carfilzomib; Etoposide; Ifosfamide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carfilzomib, rituximab, chemotherapy) (Experimental): Patients receive carfilzomib IV over 10-30 minutes on days 1, 2, 8, and 9; rituximab IV over 3-8 hours on day 3; etoposide IV over 1 hour on days 4-6; carboplatin IV over 1 hour on day 5; and ifosfamide IV over 24 hours on day 5. Treatment repeats every 21-28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Carfilzomib; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Rituximab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of carfilzomib when given together with rituximab, ifosfamide, carboplatin, and etoposide and to see how well it works in treating patients with stage I-IV diffuse large B-cell lymphoma that has returned (relapsed) or that has not responded to treatment (refractory). Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as ifosfamide, carboplatin, and etoposide, also work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving carfilzomib with rituximab, ifosfamide, carboplatin, and etoposide may be a better treatment for diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* I. To estimate the maximum tolerated dose (MTD) and examine the dose-limiting toxicities of carfilzomib when administered in combination with rituximab, ifosfamide, carboplatin, and etoposide (C-R-ICE) in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). (Phase I)
* II. To assess the toxicity of dose regimen using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0). (Phase I)
* III. To evaluate the safety of carfilzomib (given at maximum tolerated dose [MTD] as determined in Phase I of this study) in combination with R-ICE salvage therapy in relapsed/refractory DLBCL patients. (Phase Ib)
* IV. To achieve an overall response rate (complete response [CR] and partial response [PR]) of 70% after 3 cycles of C-R-ICE in patients between the ages of 18 to 75 with relapsed/refractory cluster of differentiation (CD)20-positive DLBCL previously treated with rituximab-based immunochemotherapy (e.g., rituximab, cyclophosphamide, doxorubicin, vincristine [vincristine sulfate], and prednisone [R-CHOP], rituximab, etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin [REPOCH], rituximab, cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, and cytarabine [R-HyperCVAD], etc.) induction. (Phase Ib)

SECONDARY OBJECTIVES:

* I. To determine the feasibility of successful mobilization of autologous stem cells (i.e., minimum of 2 x 10^6 CD34+ cells/kg should be collected) to be used for autologous stem cell transplant (ASCT)
* II. To determine toxicities associated with C-R-ICE salvage therapy
* III. To determine the time to progression (TTP), progression-free survival (PFS), and overall survival (OS) followed by ASCT; disease-free survival in CR patients.
* IV. To determine the pharmacokinetics/pharmacodynamics relationship between carfilzomib's degree of proteasome inhibition and response rate along with the time course of thrombocytopenia
* V. To study differences in clinical outcomes between germinal center B-cell-like (GCB) and non-GCB relapsed/refractory DLBCL following therapy with carfilzomib and R-ICE
* VI. Correlative translational research studies to include: phenotypic/genotypic analysis and functional activity (i.e., antibody-dependent cellular cytotoxicity [ADCC] and complement-mediated cytotoxicity [CMC]) of patient's peripheral blood mononuclear "effector" cells (PBMC), as well as ex vivo analysis of sensitivity of primary tumor cells to various combinations of carfilzomib versus bortezomib +/- rituximab; enzymatic assay for chymotrypsin-like activity to determine the degree of proteasome inhibition in primary DLBCL patient samples and patient PBMC specimens; explorative analysis to identify potential factors predictive of response to therapy will be performed.

OUTLINE: This is a phase I, dose-escalation study of carfilzomib, followed by a phase Ib study.

Patients receive carfilzomib intravenously (IV) over 10-30 minutes on days 1, 2, 8, and 9; rituximab IV over 3-8 hours on day 3; etoposide IV over 1 hour on days 4-6; carboplatin IV over 1 hour on day 5; and ifosfamide IV over 24 hours on day 5. Treatment repeats every 21-28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of relapsed/refractory CD20 positive diffuse large B-cell lymphoma
* Ann Arbor stage I to stage IV DLBCL at the time of relapsed/refractory disease to be eligible
* Measurable or assessable disease is required; measurable tumor size (at least one node measuring 2.25 cm^2 in bidimensional measurement) per computed tomography (CT) scan, other radiological study, and/or physical exam
* Patients must have received at least 1 prior rituximab-based immunochemotherapy (e.g., R-CHOP, R-EPOCH, etc.)
* >= 2 weeks since major surgery
* Patients must not have any significant toxicity associated with prior surgery, radiation therapy, chemotherapy, or immunotherapy, per principal investigator (PI) discretion
* Life expectancy >= 3 months
* Karnofsky score (KS) >= 50
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 3.5 times the upper limit of normal within 14 days prior to starting therapy
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L within 14 days prior to starting therapy*
* Hemoglobin >= 8 g/dL (80 g/L) within 14 days prior to randomization (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines)*
* Platelet count >= 50 x 10^9/L (>= 20 x 10^9/L if lymphoma involvement in the pretreatment bone marrow is found) within 14 days prior to starting therapy*
* *Note: If patient has cytopenias due to bone marrow involvement, these requirements are not applicable
* Serum creatinine of =< 1.5 mg/dL; if creatinine > 1.5 mg/dL creatinine clearance must be > 60 mL/min within 7 days prior to treatment either measured or calculated using a standard Cockcroft and Gault formula
* Written informed consent in accordance with federal, local, and institutional guidelines
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male subjects must agree to practice contraception
* No known hypersensitivity to murine products
* Patients must have normal baseline cardiac function based upon echocardiogram or gated blood pool scan (multigated acquisition scan [MUGA]) with an ejection fraction >= 50%
* Patients who test positive for hepatitis C (HepC) antibodies (Ab) are eligible provided all of the following criteria are met: bilirubin =< 2 x upper limit of normal; ALT/AST =< 3 x upper limit of normal; and clinical evaluation to rule out cirrhosis
* Specific guidelines will be followed regarding inclusion of relapsed/refractory DLBCL based on hepatitis B serological testing as follows:

  * Hepatitis B surface antigen (HBsAg) negative, hepatitis B core antibody (HBcAb) negative, hepatitis B surface antibody (HBsAb) positive patients are eligible
  * Patients who test positive for HBsAg are ineligible (regardless of other hepatitis B serologies)
  * Patients with HBsAg negative, but HBcAb positive (regardless of HBsAb status) should have a hepatitis B virus (HBV) deoxyribonucleic acid (DNA) testing done and protocol eligibility determined as follows:

    * If HBV DNA is positive, the subject will be excluded from the study
    * If HBV DNA is negative, the subject may be included but must undergo at least every 2 months HBV DNA polymerase chain reaction (PCR) testing from the start of treatment throughout the duration the treatment course

Exclusion Criteria:

* Patients with non-Hodgkin lymphoma (NHL) other than DLBCL; including "transformed" DLBCL
* Known to be seropositive for human immunodeficiency virus (HIV); an HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk
* Positive serology for HBV defined as a positive test for HBsAg; in addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HepB DNA test will be performed and if positive the subject will be excluded
* Patients with symptomatic brain involvement
* Peripheral neuropathy of grade 2 or greater severity as defined by the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0; patients with grade 2 or higher (NCI-Common Toxicity Criteria [CTC]) neuropathy
* Myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemia
* Uncontrolled intercurrent illness including, but not limited to, active infection, poorly controlled hypertension, diabetes mellitus or other serious medical or psychiatric conditions that could interfere with adherence to or completion of this study
* Pregnant or breastfeeding
* Patient has received other investigational drugs within 4 weeks before enrollment
* Chemotherapy within 3 weeks of the first scheduled study treatment
* Less than 2-years disease free from another primary malignancy (other than squamous or basal cell carcinoma of the skin, "in-situ" carcinoma of the cervix or breast, superficial bladder carcinoma, or previously treated localized prostate cancer with normal prostate-specific antigen [PSA] levels); patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, are considered by their physician to be at less than 30% risk of relapse and at least 2 years have lapsed
* Major surgery, other than diagnostic surgery, within 2 weeks
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Medical condition requiring chronic use of high dose systemic corticosteroids (i.e., doses of prednisone higher than 10 mg/day or equivalent)
* Prior high-dose chemotherapy (HDC)-ASCT
* Active central nervous system (CNS) disease defined as symptomatic meningeal lymphoma or known CNS parenchymal lymphoma; a lumbar puncture demonstrating DLBCL at the time of registration to this study is not exclusion for study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Hernandez-ILizaliturri, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Lin LH, Ghasemi M, Burke SM, Mavis CK, Nichols JR, Torka P, Mager DE, Hernandez-Ilizaliturri FJ, Goey AKL. Population Pharmacokinetics and Pharmacodynamics of Carfilzomib in Combination with Rituximab, Ifosfamide, Carboplatin, and Etoposide in Adult Patients with Relapsed/Refractory Diffuse Large B Cell Lymphoma. Target Oncol. 2023 Sep;18(5):685-695. doi: 10.1007/s11523-023-00992-4. Epub 2023 Aug 26. PMID 37632592

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Carfilzomib 10mg/m2 (d1-2; d8-9): Patients receive carfilzomib IV over 10-30 minutes on days 1, 2, 8, and 9; rituximab IV over 3-8 hours on day 3; etoposide IV over 1 hour on days 4-6; carboplatin IV over 1 hour on day 5; and ifosfamide IV over 24 hours on day 5. Treatment repeats every 21-28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Carfilzomib: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Rituximab: Given IV
- Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9); Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9); Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9); Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9); Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9); Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9): Patients receive carfilzomib IV over 10-30 minutes on days 1, 2, 8, and 9; rituximab IV over 3-8 hours on day 3; etoposide IV over 1 hour on days 4-6; carboplatin IV over 1 hour on day 5; and ifosfamide IV over 24 hours on day 5. Treatment repeats every 21-28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1: Carfilzomib 10mg/m2 (d1-2; d8-9) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9)
Started | 3 | 3 | 3 | 3 | 3 | 6 | 8
Completed | 2 | 3 | 2 | 1 | 3 | 3 | 4
Not Completed | 1 | 0 | 1 | 2 | 0 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 2 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9)(Carfilzomib, Rituximab, Chemotherapy); Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9); Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9); Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9); Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9); Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9); Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9): Patients receive carfilzomib IV over 10-30 minutes on days 1, 2, 8, and 9; rituximab IV over 3-8 hours on day 3; etoposide IV over 1 hour on days 4-6; carboplatin IV over 1 hour on day 5; and ifosfamide IV over 24 hours on day 5. Treatment repeats every 21-28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Carfilzomib: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Rituximab: Given IV
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9)(Carfilzomib, Rituximab, Chemotherapy) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 2 | 3 | 4 | 6 | 20
  >=65 years | 2 | 1 | 1 | 1 | 0 | 2 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (11.2) | 62.5 (4.4) | 64.6 (8.6) | 45.5 (21.3) | 58.9 (1.7) | 63.3 (4.3) | 59.1 (11.8) | 60.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 0 | 3 | 5 | 11
  Male | 1 | 3 | 2 | 3 | 3 | 3 | 3 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (PR + CR)
Description: Overall response rate (CR and PR) after 3 cycles of C R ICE in patients age of 18 to 75 with relapsed/refractory CD20-positive DLBCL treated with rituximab-based immunochemotherapy (e.g., R-CHOP, R-EPOCH, R-HyperCVAD, etc.) induction. Response was based on a Modified Cheson Criteria with Complete response (CR): All lesions with a longest diameter ≤ 15 mm or short axis ≤ 10 mm (Not palpable during the clinical examination, No visible nodule on imaging, And disappearance of all non-nodal target lesions Or in case of hypermetabolic disease on the baseline PET scan, negative PET scan whatever the appearance of lesions on CT) and Partial Response (PR): ≥ 50 % of sum of the products of the diameters (SPD) of target lesions or in the case of hypermetabolic lesions on the baseline PET scan, persistence of at least one PET-positive site without progression of other lesions on CT (≥ 50 % of SPD of target lesions (or longest diameter if a single nodule) No clinically enlarged liver or spleen)
Time Frame: The time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented, assessed up to 12 weeks
Population: All treated and eligible patients. Per the protocol "The efficacy analysis will include evaluable patients in Phase I and Phase Ib portions combined".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 29
percentage of participants | 66 [46 to 82]

2. Primary Outcome: MTD Defined as the Dose of Carfilzomib Added to Standard R-ICE Chemotherapy Which, if Exceeded, Would Put the Patient at an Undesirable Risk of Medically Unacceptable Dose-limiting Toxicities (Phase I)
Time Frame: 28 days
Population: All treated and eligible patients
Measure: Number; unit: mg/m2
Groups:
- Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9): Patients receive carfilzomib IV over 10-30 minutes on days 1, 2, 8, and 9; rituximab IV over 3-8 hours on day 3; etoposide IV over 1 hour on days 4-6; carboplatin IV over 1 hour on day 5; and ifosfamide IV over 24 hours on day 5. Treatment repeats every 21-28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Carfilzomib: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Rituximab: Given IV
Arm/Group | Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8
mg/m2 | NA — MTD was not reached. | NA — MTD was not reached. | NA — MTD was not reached. | NA — MTD was not reached. | NA — MTD was not reached. | NA — MTD was not reached. | NA — MTD was not reached.

3. Secondary Outcome: Complete Response Rate According to the International Working Group Response Criteria as Reported by the Revised Cheson Criteria
Description: Efficacy rates were estimated using simple relative frequencies. Complete response rate after 3 cycles of C R ICE in patients age of 18 to 75 with relapsed/refractory CD20-positive DLBCL treated with rituximab-based immunochemotherapy (e.g., R-CHOP, R-EPOCH, R-HyperCVAD, etc.) induction. Response was based on a Modified Cheson Criteria with Complete response (CR): All lesions with a longest diameter ≤ 15 mm or short axis ≤ 10 mm (Not palpable during the clinical examination, No visible nodule on imaging, And disappearance of all non-nodal target lesions Or in case of hypermetabolic disease on the baseline PET scan, negative PET scan whatever the appearance of lesions on CT) and Partial Response (PR): ≥ 50 % of sum of the products of the diameters (SPD) of target lesions or in the case of hypermetabolic lesions on the baseline PET scan, persistence of at least one PET-positive site without progression of other lesions on CT (≥ 50 % of SPD of target lesions (or longest diameter if a si
Time Frame: Up to 5 years
Population: All treated and eligible patients, Per the protocol "The efficacy analysis will include evaluable patients in Phase I and Phase Ib portions combined".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 29
percentage of participants | 48 [29 to 67]

4. Secondary Outcome: Overall Survival
Description: The estimated distributions of overall survival will be obtained using the Kaplan-Meier method. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed. It is assumed a priori that any drop out times will be non-informative in terms of the censoring mechanism. Groups defined by levels of categorical or dichotomized numeric demographic/baseline variables will be compared in regards to time-to-event distributions using the log-rank test. Cox proportional hazards model regression will be utilized for multivariate analyses.
Time Frame: From the start of treatment until death for any reason, assessed up to 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 29
months | 22.6 [6.6 to NA] — The upper limit was not reached. Per the protocol "The efficacy analysis will include evaluable patients in Phase I and Phase Ib portions combined".

5. Secondary Outcome: Pharmacokinetics (PK)/Pharmacodynamics (PD) of Carfilzomib and Standard R-ICE Combination Therapy in Adult Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Description: A population PK/PD structural model will be developed for carfilzomib based on degree of proteasome inhibition in relation to efficacy and toxicity endpoints in the proposed study using NONMEM. This model will describe the potential relationship between carfilzomib exposure in relation to proteasome inhibition to the time course of thrombocytopenia and neutropenia as indicators of pharmacodynamics response.
Time Frame: Pre-dose, just prior to the end of the infusion; and at 15 minutes, 30 minutes, 1, 2, 4, 6 hours post infusion on course 1, day 1, then at 24 hours post course 1 infusion on course 1, day 2 (prior to day 2 infusion)
Population: The analysis of this endpoint was contingent on ancillary grant funding, which did not occur. Hence these endpoints were not collected.
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival
Description: The estimated distributions of progression-free survival will be obtained using the Kaplan-Meier method. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed. It is assumed a priori that any drop out times will be non-informative in terms of the censoring mechanism. Groups defined by levels of categorical or dichotomized numeric demographic/baseline variables will be compared in regards to time-to-event distributions using the log-rank test. Cox proportional hazards model regression will be utilized for multivariate analyses.
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 29
months | 15.2 [5.1 to NA] — The upper limit was not reached.

7. Secondary Outcome: Toxicity of the Addition of Carfilzomib to R-ICE at the MTD, Assessed by the CTEP Version 4.0 of the NCI CTCAE
Description: Count of participants that experienced serious adverse events assessed by the CTEP version 4.0 of the NCI CTCAE
Time Frame: Up to 5 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 8
Participants | 2 | 0 | 0 | 1 | 1 | 3 | 4

8. Other Pre Specified Outcome: Degree of Proteasome Inhibition Determined by Enzymatic Assay for Chymotrypsin-like Activity
Time Frame: Days 1-3 of course 1
Population: as for outcome 5
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Ex Vivo Analysis of Sensitivity of Primary Tumor Cells to Various Combinations of Carfilzomib Versus Bortezomib +/- Rituximab
Time Frame: Baseline
Population: as for outcome 5
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Functional Activity of Patients Peripheral Blood Mononuclear "Effector" Cells
Time Frame: Baseline
Population: as for outcome 5
Arm/Group | Treatment (Carfilzomib, Rituximab, Chemotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline, weekly until 30 days after the last intervention or until the event has resolved, stabilized, death, or a new treatment is started, whichever comes first, will be reported.
Description: Assess the toxicity of dose regimen using the CTEP NCI Common Terminology Criteria for Adverse Events (CTCAE Version 4.0).
Arm/Group | Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9)
All-Cause Mortality (participants affected / at risk) | 3/3 | 0/3 | 1/3 | 3/3 | 1/3 | 4/6 | 2/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 0/3 | 1/3 | 1/3 | 3/6 | 4/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9) (N=3) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) (N=3) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) (N=3) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) (N=3) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) (N=3) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) (N=6) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Lymph node abscess (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: Carfilzomib 10mg/m2(d1-2; d8-9) (N=3) | Dose Level 2: Carfilzomib 15mg/m2(d1-2; d8-9) (N=3) | Dose Level 3: Carfilzomib 20mg/m2(d1-2; d8-9) (N=3) | Dose Level 4: Carfilzomib 20mg/m2(d1-2); 27mg/m2(d8-9) (N=3) | Dose Level 5: Carfilzomib 20mg/m2(d1-2); 36mg/m2(d8-9) (N=3) | Dose Level 6: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) (N=6) | Expansion Cohort: Carfilzomib 20mg/m2(d1-2); 45mg/m2(d8-9) (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (30) | 3 (27) | 1 (3) | 2 (9) | 2 (6) | 4 (15) | 1 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Vision blurred (Eye disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (9) | 1 (3) | 1 (3) | 2 (6) | 4 (18) | 4 (12)
Diarrhoea (Gastrointestinal disorders) | 1 (9) | 2 (6) | 2 (6) | 2 (6) | 1 (3) | 2 (9) | 2 (6)
Dry mouth (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (6) | 2 (9) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Nausea (Gastrointestinal disorders) | 2 (6) | 3 (18) | 3 (12) | 2 (9) | 2 (6) | 4 (15) | 4 (15)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 3 (9) | 3 (9) | 0 (0) | 1 (3) | 1 (3) | 2 (6) | 0 (0)
Asthenia (General disorders) | 3 (9) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (6) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Extravasation (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (12) | 0 (0) | 2 (6) | 3 (9) | 3 (9) | 2 (6) | 3 (9)
Infusion site erythema (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 2 (6) | 1 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (3) | 1 (3) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 2 (6)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (21) | 3 (24) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 2 (6)
Platelet count decreased (Investigations) | 3 (24) | 3 (21) | 1 (3) | 3 (21) | 2 (6) | 5 (18) | 4 (15)
Prothrombin time prolonged (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (9) | 2 (21) | 1 (3) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 2 (6) | 2 (6) | 1 (3) | 2 (9) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (24) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 2 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (6) | 2 (6) | 0 (0) | 1 (3) | 1 (3) | 1 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (9) | 1 (3) | 2 (6) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (3) | 1 (3) | 2 (6) | 2 (6) | 0 (0) | 2 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (6) | 0 (0) | 2 (9) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (12) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (3) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (6) | 2 (6) | 1 (3) | 2 (6) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (6) | 2 (9) | 1 (3) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 3 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (9) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 4 (12) | 4 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Hypotension (Vascular disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT01959698/Prot_SAP_000.pdf